CLINICAL TRIAL: NCT06688539
Title: A Prospective Trial of Varenicline and Incentives for E-cigarette Cessation in Adults Who Co-use Cannabis
Brief Title: E-cigarette Cessation in Adults Who Co-use Cannabis
Acronym: VapeCAT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Erin McClure, Associate Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00136601; R37CA237245 (NIH)
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2025-07-07 (Actual); Status verified 2025-07

CONDITIONS: Nicotine Dependence; Tobacco Use Disorder
Keywords: e-cigarettes; cannabis; treatment
MeSH Terms: conditions — Tobacco Use Disorder; Vaping; Marijuana Abuse | interventions — Varenicline; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Co-use group (Other): E-cigarette and cannabis co-use group
  Interventions: Drug: Varenicline Pill; Behavioral: Contingency management; Behavioral: Counseling

INTERVENTIONS:
Drug: Varenicline Pill — In this study, all participants will be administered active medication for a 12 week treatment period. The standard dose titration schedule will be used, which includes 0.5 mg once per day (q.d.) on Days 1-3, 0.5 mg twice per day (b.i.d.) on Days 4-7, and 1.0 mg b.i.d. starting on Day 8. Dosing of 2.0 mg per day will be maintained for the next 11 weeks, for a total of 12 weeks of active treatment for all study participants.
Behavioral: Contingency management — Contingency management procedures will be implemented and financial incentives will be provided at weekly visits contingent on e-cigarette abstinence verified through urinary qualitative cotinine (starting at Week 2). A set amount of $20 per study visit will be delivered based on a negative qualitative urinary cotinine result.
Behavioral: Counseling — Psychosocial counseling will be administered by trained research staff leading up to the target quit date and throughout the study.

SUMMARY:
The purpose of this study is to better understand tobacco outcomes using a commonly prescribed stop smoking medication (varenicline) and financial incentives for adults who also use cannabis. Varenicline is not FDA approved for e-cigarette cessation, but is FDA approved for cigarette cessation. Investigators are also interested in how cannabis/marijuana and tobacco interact during a tobacco quit attempt. All participants will receive e-cigarette cessation treatment for 12 weeks. To qualify, participants must be between the ages of 18-40 and use both e-cigarettes and cannabis. Participants do not need to be interested in quitting cannabis to qualify. This study is being conducted at three sites: the Medical University of South Carolina in Charleston, SC, Behavioral Health Services in Pickens, SC, and MUSC Lancaster in Lancaster, SC.

DETAILED DESCRIPTION:
Cannabis co-use among tobacco users is exceedingly common and rates of co-use appear to be increasing among adults in the US, which is consistent with overall increases in cannabis use rates among US adults. Given the current cannabis landscape, further increases in cannabis use are likely and may result in continued increases in the co-use of cannabis and tobacco.

Despite high rates of co-use, there is little consensus regarding treatment recommendations for this population and an understanding of the impact of co-use on successful cessation. The literature on the impact of co-use on tobacco cessation outcomes specifically has been mixed and fraught with limitations, including methodological variation, lack of biochemical verification to confirm cannabis use status and severity, and variations in study samples. Currently, no prospective studies have been conducted to evaluate the impact of cannabis use on tobacco cessation outcomes. Further, no studies have collected cannabis use changes during tobacco cessation treatment to assess for concurrent reductions, abstinence, or of greater concern, compensatory (i.e., increased) use as a result of tobacco reduction/abstinence.

This study is a prospective 12-week tobacco cessation trial using established methods and outcomes typical of tobacco cessation trials, but specifically recruiting co-users of cannabis. The aims of this proposed study are to; Specific Aim 1. Compare rates of 7-day biochemically-confirmed e-cigarette abstinence with cigarette abstinence rates from the parent R37 co-use sample (as a historical controls). Specific Aim 2. Assess changes in cannabis use during e-cigarette cessation treatment among the new sample of participants enrolled in this extension.

Specific Aim 3. Assess for a dose-dependent impact of cannabis co-use severity on e-cigarette cessation. Specific Aim 4. Characterize and compare patterns of co-use among the e-cigarette sample to those using cigarettes (parent R37).

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 40 years old
* Use e-cigarettes daily or near daily in the past month
* Must submit a positive instant-read urine cotinine test at screening (≥ 200 ng/ml)
* Be interested in quitting use of e-cigarettes
* Must be willing to take varenicline for the standard 12-week course of treatment
* Self-reported use of cannabis on at least 10 out of the past 30 days or must submit a positive qualitative urinary cannabinoid test at screening (> 50 ng/ml)

Exclusion Criteria:

* Any serious or unstable medical/psychiatric disorder (including severe substance use disorders, other than cannabis or tobacco use disorders) in the past three months that may interfere with study performance
* Use of cigarettes on 10+ days in the past 30
* Currently pregnant or breastfeeding
* Current use of medications with smoking cessation efficacy
* Use of any medications that would interfere with varenicline

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-02-19 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
7-day point prevalence tobacco abstinence at the end of treatment (Week 12) | Final 7 days of treatment (Week 12)
  7-day point prevalence abstinence from e-cigarettes at the end of treatment (Week 12) will be assessed via biochemical verification (urinary cotinine; ng/ml) and will be compared to cigarette abstinence rates from the parent study (as historical controls)

SECONDARY OUTCOMES:
Changes in cannabis use during e-cigarette cessation treatment | Final 4 weeks of study treatment (Weeks 8-12)
  Cannabis use rates (based on urinary cannabinoids [ng/ml]) during the final 4 weeks of tobacco treatment (Weeks 8-12) will be assessed.
Cannabis co-use severity on e-cigarette abstinence rates | Final 7 days of treatment (Week 12)
  Assess for a dose-dependent impact of cannabis co-use severity on e-cigarette cessation.

CONTACTS AND LOCATIONS:
Overall Officials: Erin A McClure, PhD, Principal Investigator — Medical University of South Carolina
Locations (3):
- United States (3):
  - MUSC Charleston, Charleston, South Carolina
  - MUSC Lancaster, Lancaster, South Carolina
  - Behavioral Health Services of Pickens County, Pickens, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available for retrieval and analysis of secondary outcomes, upon request to the Principal Investigator. Study datasets (de-i
Supporting Information: Study Protocol, ICF